CLINICAL TRIAL: NCT04284150
Title: Treatment of Supraventricular Tachycardia in Patients With Non-cardiac Surgery by Dexmedetomidine During the Perioperative Period
Brief Title: Treatment of Supraventricular Tachycardia in Patients With Non-cardiac Surgery by Dexmedetomidine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lianyungang Hospital Affiliated Bengbu Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019101201
Record Dates: First submitted 2020-02-13; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Perioperative Period
Keywords: Supraventricular tachycardia; Dexmedetomidine; Midazolam; Heart rate variability
MeSH Terms: conditions — Tachycardia, Supraventricular | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Intervention Model Description: patients with supraventricular tachycardia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dexmedetomidine or Midazola treat supraventricular tachycardia (Experimental): Comparison of efficacy of dexmedetomidine and Midazolam in the treatment of SVT
  Interventions: Drug: Dexmedetomidine; Midazolam;

INTERVENTIONS:
Drug: Dexmedetomidine; Midazolam; — Treatment of supraventricular tachycardia in patients with non-cardiac surgery by dexmedetomidine during the perioperative period
  Other Names: supraventricular tachycardia

SUMMARY:
Supraventricular tachycardia (SVT) is a common arrhythmia in the perioperative period, which is associated with adverse stimulus such as cardiovascular risk factors, emotional tension, hypoxia, CO2 accumulation, hypokalemia, atropine and pain. To treat perioperative SVT, in addition to massage the vagus nerve, the use of antiarrhythmic drugs and other internal medicine classic methods, the cardiovascular protection of anesthetic drugs is also a common adjuvant treatment. Dexmedetomidine which is widely used as an adjuvant to general anesthesia, can excite α2 receptor to produce sedation, analgesia, inhibition of sympathetic activity, stabilization of hemodynamics and other effects.

Dexmedetomidine is approved by FDA for use in operating room anesthesia and intensive care unit sedation in adults. Although dexmedetomidine is not approved for the treatment of arrhythmias, a growing number of evidences indicated dexmedetomidine can serve as a potential treatment for arrhythmias in perioperative patients. Liu et al. confirmed that dexmedetomidine can reduce ventricular rate and improve atrial fibrillation in cardiac surgery patient. Ji et al. showed that dexmedetomidine anesthesia can be effective in lowering cardiovascular and cerebrovascular complications and mortality in patients one year after coronary bypass surgery. A number of retrospective analyses of pediatric patients undergoing cardiac surgery have shown the incidence of perioperative SVT in patients treated with dexmedetomidine sedation is significantly decreased, which prompts that dexmedetomidine has the potential prevention and treatment for tachyarrhythmia. Therefore, the investigators selected dexmedetomidine for sedation in patients with perioperative SVT to explore the effect for treating SVT via its sedation and mechanism of anti-sympatheticon in this study.

DETAILED DESCRIPTION:
Forty patients with SVT of both sexes, aged 35-61 yr, of American Society of Anesthesiologists physical status Ⅰ-Ⅱ, who undergo elective surgery, were randomly divided into two groups (n=30) including dexmedetomidine group (group D) and midazolam group (group M). For comparison of the efficacy of dexmedetomidine and midazolam in the treatment of SVT, the following needs to be done. The patients calm down for 5-10 minutes after getting into the operating room, group D and group M started as a continuous infusion with dexmedetomidine 0.5µg/kg or midazolam 0.06mg/kg using a micro-pump for 10 minutes. The alarm/sedation (OAA/S) score, heart rate (HR), mean arterial pressure (MAP), pulse oxygen saturation (SpO2) and occurrence of SVT were recorded before the infusion (T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4). In two groups, miniature electrocardiograph was used to monitor the frequency domain index of heart rate variability (HRV) in 5 minutes at each time point including normalized low frequency power (LFnorm), normalized high frequency power (HFnorm) and the balance ratio of sympathetic to vagal tone (LF/HF).

ELIGIBILITY:
Inclusion Criteria:

* Patients with supraventricular tachycardia

Exclusion Criteria:

* Patients who suffered from significant hemodynamic instability, and can not receive dexmedetomidine and midazolam, were thus excluded from the study.
* Patients with other types of arrhythmia, not SVT, abnormal liver and kidney function and anaesthesia-related drug allergy, were excluded from the study.

Ages: 35 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-26 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
dexmedetomidine treat supraventricular tachycardia | through study completion, up to 6 months
  effective rate of dexmedetomidine on supraventricular tachycardia
midazolam treat supraventricular tachycardia | through study completion, up to 6 months
  effective rate of midazolam on supraventricular tachycardia
Comparison of efficacy of dexmedetomidine and midazolam in the treatment of SVT | through study completion, up to 6 months
  occurrence of SVT recorded before the infusion dexmedetomidine and midazolam (T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4) in two groups

SECONDARY OUTCOMES:
alarm/sedation (OAA/S) score | through study completion, up to 6 months
  This indicator was recorded before the infusion dexmedetomidine and midazolam(T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4) in two groups for evaluating the efficacy of dexmedetomidine and midazolam in the treatment of SVT
heart rate (HR) | through study completion, up to 6 months
  This indicator was recorded before the infusion dexmedetomidine and midazolam(T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4) in two groups for evaluating the efficacy of dexmedetomidine and midazolam in the treatment of SVT
mean arterial pressure (MAP) | through study completion, up to 6 months
  This indicator was recorded before the infusion dexmedetomidine and midazolam(T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4) in two groups for evaluating the efficacy of dexmedetomidine and midazolam in the treatment of SVT
pulse oxygen saturation (SpO2) | through study completion, up to 6 months
  This indicator was recorded before the infusion dexmedetomidine and midazolam(T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4) in two groups for evaluating the efficacy of dexmedetomidine and midazolam in the treatment of SVT
normalized low frequency power | through study completion, up to 6 months
  This indicator was recorded before the infusion dexmedetomidine and midazolam(T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4) in two groups for evaluating the efficacy of dexmedetomidine and midazolam in the treatment of SVT
normalized high frequency power | through study completion, up to 6 months
  This indicator was recorded before the infusion dexmedetomidine and midazolam(T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4) in two groups for evaluating the efficacy of dexmedetomidine and midazolam in the treatment of SVT
the balance ratio of sympathetic to vagal tone | through study completion, up to 6 months
  This indicator was recorded before the infusion dexmedetomidine and midazolam(T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4) in two groups for evaluating the efficacy of dexmedetomidine and midazolam in the treatment of SVT This indicator was recorded before the infusion dexmedetomidine and midazolam(T0), 5 minutes after the infusion (T1), at the end of the infusion (T2), 5 minutes after the end of the infusion (T3) and 10 minutes after the end of the infusion (T4) in two groups for evaluating the efficacy of dexmedetomidine and midazolam in the treatment of SVT

CONTACTS AND LOCATIONS:
Overall Officials: Junlong Zhang, PhD, Principal Investigator — the Affiliated Lianyungang No. 2 People's Hospital of Jiangsu University

REFERENCES:
- [Result] Alabed S, Sabouni A, Providencia R, Atallah E, Qintar M, Chico TJ. Adenosine versus intravenous calcium channel antagonists for supraventricular tachycardia. Cochrane Database Syst Rev. 2017 Oct 12;10(10):CD005154. doi: 10.1002/14651858.CD005154.pub4. PMID 29025197
- [Result] Zhu SJ, Wang KR, Zhang XX, Zhu SM. Relationship between genetic variation in the alpha2A-adrenergic receptor and the cardiovascular effects of dexmedetomidine in the Chinese Han population. J Zhejiang Univ Sci B. 2019 Jul;20(7):598-604. doi: 10.1631/jzus.B1800647. PMID 31168973
- [Result] Black N, D'Souza A, Wang Y, Piggins H, Dobrzynski H, Morris G, Boyett MR. Circadian rhythm of cardiac electrophysiology, arrhythmogenesis, and the underlying mechanisms. Heart Rhythm. 2019 Feb;16(2):298-307. doi: 10.1016/j.hrthm.2018.08.026. Epub 2018 Aug 29. PMID 30170229
- [Result] Jung W, Jang KI, Lee SH. Heart and Brain Interaction of Psychiatric Illness: A Review Focused on Heart Rate Variability, Cognitive Function, and Quantitative Electroencephalography. Clin Psychopharmacol Neurosci. 2019 Nov 20;17(4):459-474. doi: 10.9758/cpn.2019.17.4.459. PMID 31671483
- [Result] Chrysostomou C, Morell VO, Wearden P, Sanchez-de-Toledo J, Jooste EH, Beerman L. Dexmedetomidine: therapeutic use for the termination of reentrant supraventricular tachycardia. Congenit Heart Dis. 2013 Jan-Feb;8(1):48-56. doi: 10.1111/j.1747-0803.2012.00669.x. Epub 2012 May 22. PMID 22613357
- [Result] Liu X, Zhang K, Wang W, Xie G, Fang X. Dexmedetomidine sedation reduces atrial fibrillation after cardiac surgery compared to propofol: a randomized controlled trial. Crit Care. 2016 Sep 21;20(1):298. doi: 10.1186/s13054-016-1480-5. PMID 27654700